CLINICAL TRIAL: NCT03466866
Title: Randomized Controlled Trial of Preventing and Reducing Emergency Visits in Diabetes Through Education and Telehealth vs. Diabetes Education to Reduce Emergency Visits and Hospitalizations Over 12 Months in African Americans Americans
Brief Title: Reducing Emergency Diabetes Care for Older African Americans
Acronym: PREVENT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Barry Rovner, PI, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: R01DK114033-01A1 (NIH)
Record Dates: First submitted 2018-03-09; First posted 2018-03-15 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Single blind, randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PREVENT (Preventing and Reducing Emergency Visits in Diabetes through Education and Telehealth) (Experimental): Community Health Workers (CHWs), who are race-concordant with participants, will: 1) deliver in-home DM education to increase participants' knowledge and skills; 2) use DM-specific Behavioral Activation to improve DM self-care; and 3) facilitate telehealth visits with the participant's primary care physician (PCP) and a DM nurse educator to increase access to care.
  Interventions: Behavioral: PREVENT
- EUC (Enhanced Usual Care) (Active Comparator): In-home diabetes education with no goal setting or telehealth visits
  Interventions: Behavioral: EUC (Enhanced Usual Care)

INTERVENTIONS:
Behavioral: PREVENT — Community Health Workers (CHWs), who are race-concordant with participants, will: 1) deliver in-home DM education to increase participants' knowledge and skills; 2) use DM-specific Behavioral Activation to improve DM self-care; and 3) facilitate telehealth visits with the participant's primary care physician (PCP) and a DM nurse educator to increase access to care.
  Other Names: COPDE (former name)
  Arms: PREVENT (Preventing and Reducing Emergency Visits in Diabetes through Education and Telehealth)
Behavioral: EUC (Enhanced Usual Care) — In-home diabetes education with no goal setting or telehealth visits
  Arms: EUC (Enhanced Usual Care)

SUMMARY:
This RCT will compare the efficacy of Preventing and Reducing Emergency Visits in Diabetes through Education and Trust (PREVENT) vs. intensive home-based diabetes (DM) education [i.e., Enhanced Usual Care (EUC)] to reduce DM-related emergency department (ED) visits and/or hospitalizations over 12 months (primary outcome) in 230 blacks with diabetes, 50 years and older, after an ED visit. A moderation analysis will determine whether participants who reside in low- vs. high-need communities [defined by Community Need Index scores (i.e., an indicator of the built environment)] respond differently to treatment.

PREVENT is a collaborative intervention of Primary Care Physicians, (PCPs), a DM nurse educator, and Community Health Workers (CHWs) that extends from the ED into the community. The CHWs will: 1) deliver in-home DM education to increase participants' knowledge and skills to manage DM; 2) use DM-specific Behavioral Activation to reinforce DM self-care; and 3) facilitate telehealth visits with PCPs and a DM nurse educator to increase access to care. The control treatment, EUC, is home-based intensive DM education. EUC matches PREVENT in treatment intensity (i.e., number and duration of in-home visits) and delivery of DM self-care education, but does not include PREVENTS's other active elements (i.e., Behavioral Activation and telehealth). The treatment comparison will identify PREVENTS's specific efficacy over and above EUC. We hypothesize that PREVENT will halve the rate of incident DM-related ED visits and/or hospitalizations relative to EUC. The three secondary outcomes are: 1) subjective perceptions of access to care; 2) receipt of DM Quality Metrics (i.e., objective indicators of realized access to care); and 3) DM self-care.

DETAILED DESCRIPTION:
This Phase-III RCT will compare the efficacy of Preventing and Reducing Emergency Visits in Diabetes through Education and Trust (PREVENT) vs. intensive home-based DM education to reduce the number of DM-related ED visits and/or hospitalizations over 12 months (primary outcome), in 230 AAs with DM, 40 years and older, who are recruited from the ED after an ED visit. PREVENT is a culturally relevant intervention that extends from the ED to the community, and aims to improve access to care and DM self-care (secondary outcomes). A mediation analysis will determine whether changes in access to care and/or DM self-care explain PREVENT's efficacy. A moderation analysis will determine whether participants who reside in low- vs. high-need communities [defined by Community Need Index scores (i.e., an indicator of the built environment)] respond differently to treatment.

PREVENT will begin soon after the participant's index ED visit, when many patients remain uncertain how to manage DM or how to access follow-up care. Community Health Workers (CHWs), who are race-concordant with participants, will: 1) deliver in-home DM education to increase participants' knowledge and skills; 2) use DM-specific Behavioral Activation to improve DM self-care; and 3) facilitate telehealth visits with the participant's primary care physician (PCP) and a DM nurse educator to increase access to care. The control treatment, EUC, is intensive home-based DM education. EUC matches PREVENT in treatment intensity (i.e., 6 in-home sessions over 4 months, and 3 booster sessions over the next 8 months) and delivery of culturally relevant DM education, but does not include DM-specific Behavioral Activation or telehealth visits. The treatment comparison will identify PREVENT's specific efficacy over and above EUC.

This RCT is significant as the population ages and becomes more racially diverse, and as ED use and costs increase. This RCT is innovative because it: 1) tests the first ED-to-community intervention designed to reduce the need for ED care in AAs with DM; 2) assesses both subjective and objective indicators of access to care; and 3) defines the specific characteristics of COPDE that confer its cultural relevance. If successful, PREVENT will meet Healthy People 2020's twin goals of reducing the personal and societal costs of DM and achieving health equity for all Americans. The Specific Aims of this RCT are:

Primary Specific Aim: Test the efficacy of PREVENT to reduce the number of incident DM-related ED visits and/or hospitalizations over 12 months (primary outcome) in AAs with DM. Hypothesis: PREVENT will halve the number of incident DM-related ED visits and/or hospitalizations relative to EUC over 12 months.

The Secondary Aims are to:

1. Test the efficacy of PREVENT to increase perceived access to care over 12 months (secondary outcome). Hypothesis: PREVENT will increase Patient Satisfaction Questionnaire-18 scores to a greater extent than EUC over 12 months.
2. Test the efficacy of PREVENT to increase realized access to care over 12 months (secondary outcome). Hypothesis: PREVENT will increase the number of received Diabetes Quality Metrics (e.g., hemoglobin A1c testing, urine screening) to a greater extent than EUC over 12 months.
3. Test the efficacy of PREVENT to improve DM self-care over 12 months (secondary outcome). Hypothesis: PREVENT will increase Diabetes Self-Care Inventory scores to a greater extent than EUC over 12 months.
4. Determine if increasing subjective and/or objective indicators of access to care and/or DM self-care mediates PREVENT's reduction of DM-related ED visits and/or hospitalizations. Hypothesis: PREVENT will reduce DM-related ED visits and/or hospitalizations to the extent that it increases subjective and/or objective indicators of access to care and/or improves DM self-care.

The Exploratory Aims are to: 1) determine whether PREVENT reduces "all cause" ED visits/hospitalizations relative to EUC.; 2) determine whether Community Need Index scores, literacy, age, and/or sex moderate treatment effects; 3) determine if PREVENT improves glycemic control (i.e., lowers hemoglobin A1c levels), impacts DM-related health beliefs, reduces depression, and/or improves quality-of-life; 4) identify PREVENT's treatment features that confer its cultural relevance; and 5) estimate PREVENT's costs and net financial benefit to the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

1. African American race (self-identified)
2. Age ≥ 40 years
3. Type 1 or 2 DM
4. A DM-related cause for the ED visit in the opinion of the ED physician
5. Has a Jefferson PCP (participants receiving PREVENT will have a telehealth visit with their Jefferson PCP).

Exclusion Criteria:

1. Medical or psychiatric morbidity (e.g., acute stroke, schizophrenia) that would preclude study participation in the opinion of the ED physician
2. Clinically significant cognitive impairment
3. Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry W Rovner, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 1/10/2019 to 10/13/2021
Groups:
- EUC (Enhanced Usual Care): In-home diabetes education with no goal stetting or telehealth visits
Period: Overall Study
Arm/Group | PREVENT (Preventing and Reducing Emergency Visits in Diabetes Through Education and Telehealth) | EUC (Enhanced Usual Care)
Started | 78 | 78
Completed | 62 | 62
Not Completed | 16 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PREVENT (Preventing and Reducing Emergency Visits in Diabetes Through Education and Telehealth) | EUC (Enhanced Usual Care) | Total
Number analyzed (Participants) | 78 | 78 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (9.5) | 57.2 (9.5) | 56.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 50 | 98
  Male | 30 | 28 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 77 | 76 | 153
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 78 | 78 | 156
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 78 | 78 | 156
Stratification variable: Baseline HbA1c < 9.0% vs. > or equal to 9.0% [Count of Participants; unit: Participants]
  Baseline HbA1c < 9.0% | 40 | 42 | 82
  Baseline HbA1c > or equal to 9.0% | 38 | 36 | 74
Stratification variable: Primary care physician at Jefferson [Count of Participants; unit: Participants]
  Jefferson primary care physician | 40 | 40 | 80
  Non-Jefferson primary care physician | 38 | 38 | 76
Stratification variable: Discharge status [Count of Participants; unit: Participants]
  Discharged home from index visit | 38 | 39 | 77
  Admitted from index visit | 40 | 39 | 79

OUTCOME MEASURES:

1. Primary Outcome: Number of Incident Diabetes-related ED Visits and/or Hospitalizations
Description: The primary efficacy analysis will consider the number of incident diabetes-related ED visits and/or hospitalizations (i.e., an "event") over 12 months after the index ED visit. Each ED visit or hospitalization is counted as a single event (although an ED visit that leads to a hospitalization is counted once). ED visits and hospitalization will be ascertained through chart reviews and subject self-report.
Time Frame: 12 months
Population: All randomized participants
Measure: Mean (95% Confidence Interval); unit: Incidence rate ratio
Arm/Group | PREVENT (Preventing and Reducing Emergency Visits in Diabetes Through Education and Telehealth) | EUC (Enhanced Usual Care)
Number analyzed (Participants) | 78 | 78
Incidence rate ratio | .88 [.62 to 1.27] | 1.29 [.93 to 1.79]
Statistical Analysis 1: Comparison: PREVENT (Preventing and Reducing Emergency Visits in Diabetes Through Education and Telehealth) vs EUC (Enhanced Usual Care); We used Poisson regression to model the number of outcome events as a function of randomization assignment, adjusting for the stratification variables and using follow-up time as the offset term. We calculated estimates of annual rates of the primary outcome and the adjusted estimate of the rate ratio. We evaluated the primary hypothesis by testing the null hypothesis that the rate ratio for randomization assignment equals 1; Test type: Superiority; p = .12, Poisson regression; We adjusted for stratification variables, sex, baseline MOCA, number of medical conditions, PSQ Communication, and PSQ General satisfaction; Incidence rate ratio = .67, 95% CI 2-sided [.42 to 1.07]

2. Secondary Outcome: Perceived Access to Health Care
Description: Patient Satisfaction Questionnaire scores: Mean change from baseline to 12 months. There are seven subscales, and subscale scores range from 1 to 5 with higher scores indicating greater satisfaction.
Time Frame: 12 months
Population: Participants who provided self-reported data at 6 and 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PREVENT (Preventing and Reducing Emergency Visits in Diabetes Through Education and Telehealth) | EUC (Enhanced Usual Care)
Number analyzed (Participants) | 54 | 58
units on a scale
  General Satisfaction | .22 [-.02 to .46] | .11 [-.13 to .34]
  Financial Aspects | .13 [-.12 to .39] | .29 [.04 to .55]
  Communication | .2 [-.01 to .42] | .17 [-.04 to .38]
  Accessibility and Convenience | .28 [.07 to .49] | .21 [0 to .41]
  Interpersonal Manner | .18 [-0.01 to .37] | .09 [-.09 to .28]
  Technical Quality | .27 [.07 to .46] | .17 [-.02 to .37]
  Time Spent with Doctor | .03 [-.19 to .26] | .19 [-.03 to .41]
Statistical Analysis 1: Comparison: PREVENT (Preventing and Reducing Emergency Visits in Diabetes Through Education and Telehealth) vs EUC (Enhanced Usual Care); We modeled PSQ- scores as continuous variables to estimate average change over time by treatment group. We used mixed effects linear regression with fixed effects for time (baseline, and months 6 and 12), randomization assignment, and time by randomization interaction. A random intercept term and an appropriate covariance structure was used to account for correlation among repeated measurements; Test type: Superiority — General Satisfaction; p = .502, Regression, Linear; Mean Difference (Final Values) = .11, 95% CI 2-sided [-.22 to .45]

3. Secondary Outcome: Actual Access to Care
Description: Number of received Diabetes Quality Metrics (e.g., hemoglobin A1c testing, urine screening) by 12 months. The metrics are at least 2 HbA1c tests, 1 lipid test, 1 blood pressure check, 1 diabetes foot exam, and 1 dilated fundus examination. Scores range from 0 to 6, with 6 indicating better access to care.
Time Frame: 12 months
Population: All randomized participants
Measure: Mean (95% Confidence Interval); unit: Number of quality metrics met
Arm/Group | PREVENT (Preventing and Reducing Emergency Visits in Diabetes Through Education and Telehealth) | EUC (Enhanced Usual Care)
Number analyzed (Participants) | 78 | 78
Number of quality metrics met | 3.69 [3.39 to 4.00] | 3.42 [3.12 to 3.73]
Statistical Analysis 1: Comparison: PREVENT (Preventing and Reducing Emergency Visits in Diabetes Through Education and Telehealth) vs EUC (Enhanced Usual Care); Analysis of covariance was performed with Number of Quality Metrics as the dependent variable, treatment arm as the main independent variable of interest and the stratification variables as adjusting variables; Test type: Superiority; p = .23, ANCOVA; Mean Difference (Final Values) = .26, 95% CI 2-sided [.16 to .69]

4. Secondary Outcome: Change From Baseline to 12 Months on Diabetes Self-Care Inventory Scores
Description: Frequency of engaging in diabetes self-care behaviors; Scores range from 0 to 100 with higher scores indicating more frequent engagement in diabetes self-management behaviors.
Time Frame: 12 months
Population: Participants who provided self-reported data at 6 and 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PREVENT (Preventing and Reducing Emergency Visits in Diabetes Through Education and Telehealth) | EUC (Enhanced Usual Care)
Number analyzed (Participants) | 57 | 60
units on a scale | 8.02 [4.31 to 11.73] | 3.57 [-.09 to 7.23]
Statistical Analysis 1: Comparison: PREVENT (Preventing and Reducing Emergency Visits in Diabetes Through Education and Telehealth) vs EUC (Enhanced Usual Care); We used mixed effects linear regression. Fixed effects included time (baseline, and months 6 and 12), randomization assignment, time by randomization interaction, and the three stratification variables. From the results of this model, we estimated the mean change from baseline to 6 months, 6 months to 12 months and baseline to 12 months within each treatment group. We then compared the change from baseline to 12 months between the two groups; Test type: Superiority; p = .094, Mixed Models Analysis; Mean Difference (Net) = 4.45, 95% CI 2-sided [-.76 to 9.66]

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events were events that resulted in a hospitalization. Adverse Events were reported by organ system class.
Arm/Group | PREVENT (Preventing and Reducing Emergency Visits in Diabetes Through Education and Telehealth) | EUC (Enhanced Usual Care)
All-Cause Mortality (participants affected / at risk) | 0/78 | 1/78
Serious Adverse Events (participants affected / at risk) | 36/78 | 39/78
Other Adverse Events (participants affected / at risk) | 0/78 | 0/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PREVENT (Preventing and Reducing Emergency Visits in Diabetes Through Education and Telehealth) (N=78) | EUC (Enhanced Usual Care) (N=78)
Gastrointestinal (Gastrointestinal disorders) | 5 (6) | 10 (15)
Cardiac (Cardiac disorders) | 9 (11) | 16 (22)
Diabetes-related (Endocrine disorders) | 5 (5) | 6 (6)
metabolic-not diabetes related (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Infection (Infections and infestations) | 10 (11) | 9 (14)
Stroke (Nervous system disorders) | 2 (3) | 2 (2)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
musculoskeletal (Musculoskeletal and connective tissue disorders) | 9 (13) | 5 (5)
Blood disorders (Blood and lymphatic system disorders) | 2 (7) | 3 (3)
Neurological (excluding stroke) (Nervous system disorders) | 6 (6) | 6 (7)
psychiatric (Psychiatric disorders) | 1 (1) | 1 (1)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
renal (Renal and urinary disorders) | 2 (3) | 3 (6)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7)
Surgical (Surgical and medical procedures) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT03466866/Prot_SAP_002.pdf